CLINICAL TRIAL: NCT00240331
Title: A Study to Evaluate the Use of Rosuvastatin in Subjects On Regular Haemodialysis: an Assessment of Survival and Cardiovascular Events (AURORA). A Double Blind, Randomised, Phase 3b, Parallel-group Study to Compare the Effects of Rosuvastatin With Placebo on Assessment of Survival & Cardiovascular Events When Given to Subjects With End-stage Renal Failure on Chronic Haemodialysis Treatment
Brief Title: AURORA: Crestor 10mg Versus Placebo in Subjects With End-stage Renal Disease (ESRD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: MSD, AstraZeneca
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 4522IL/0096; D3562C00096
Record Dates: First submitted 2005-10-16; First posted 2005-10-18 (Estimated); Results first posted 2009-11-04 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2011-05

CONDITIONS: Renal Failure
Keywords: End Stage Renal Failure
MeSH Terms: conditions — Renal Insufficiency; Renal Insufficiency, Chronic | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (2):
- Rosuvastatin 10mg (Experimental)
  Interventions: Drug: 10mg Rosuvastatin
- Placebo (Placebo Comparator): matching Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 10mg Rosuvastatin
  Arms: Rosuvastatin 10mg
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to see if rosuvastatin helps to reduce the number of heart attacks, strokes and cardiovascular deaths in patients undergoing haemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects with end-stage renal failure aged 50-80 years, who have received regular haemodialysis treatment for at least 3 months

Exclusion Criteria:

* Subjects will have no underlying condition that is expected to limit survival to less than 1 year and is also unrelated to end-stage renal disease (ESRD). Subjects should not have received a statin therapy within the past 6 months

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2776 (Actual)
Dates: Start 2003-01; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Crestor Medical Sciences Director, MD, Study Director — AstraZeneca
Locations (239):
- Australia (2):
  - Research Site, St Leonards, New South Wales
  - Research Site, Herston, Queensland
- Austria (8):
  - Research Site, Bregenz
  - Research Site, Feldkirch-Tisis
  - Research Site, Graz
  - Research Site, Innsbruck
  - Research Site, Linz
  - Research Site, Sankt Pölten
  - Research Site, Vienna
  - Research Site, Wels
- Belgium (6):
  - Research Site, Aalst
  - Research Site, Antwerp
  - Research Site, Brussels
  - Research Site, La Louvière
  - Research Site, Leuven
  - Research Site, Liège
- Brazil (2):
  - Research Site, Curitiba, Paraná
  - Research Site, São Paulo, São Paulo
- Bulgaria (3):
  - Research Site, Pleven
  - Research Site, Plovdiv
  - Research Site, Sofia
- Canada (19):
  - Research Site, Calgary, Alberta
  - Research Site, Edmonton, Alberta
  - Research Site, Lethbridge, Alberta
  - Research Site, Kelowna, British Columbia
  - Research Site, Vancouver, British Columbia
  - Research Site, Winnipeg, Manitoba
  - Research Site, Saint John, New Brunswick
  - Research Site, Halifax, Nova Scotia
  - Research Site, London, Ontario
  - Research Site, Mississauga, Ontario
  - Research Site, Scarborough Village, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, York, Ontario
  - Research Site, Greenfield Park, Quebec
  - Research Site, Laval, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Trois-Rivières, Quebec
  - Research Site, Kitchener
  - Research Site, Rosemount
- Czechia (7):
  - Research Site, Hodonín
  - Research Site, Hradec Králové
  - Research Site, Liberec
  - Research Site, Pardubice
  - Research Site, Prague
  - Research Site, Tábor
  - Research Site, Ústí nad Labem
- Denmark (11):
  - Research Site, Fredericia
  - Research Site, Frederiksberg
  - Research Site, Herlev
  - Research Site, Holbæk
  - Research Site, Horsens
  - Research Site, København Ø
  - Research Site, Roskilde
  - Research Site, Rønne
  - Research Site, Slagelse
  - Research Site, Sønderborg
  - Research Site, Viborg
- Finland (11):
  - Research Site, Ekenäs
  - Research Site, Helsinki
  - Research Site, Hyvinkää
  - Research Site, Joensuu
  - Research Site, Kotka
  - Research Site, Kuopio
  - Research Site, Lahti
  - Research Site, Oulu
  - Research Site, Pori
  - Research Site, Tampere
  - Research Site, Turku
- France (28):
  - Research Site, Amiens
  - Research Site, Annonay
  - Research Site, Aubervilliers
  - Research Site, Beauvais
  - Research Site, Béthune
  - Research Site, Boulogne-sur-Mer
  - Research Site, Chambéry
  - Research Site, Champigny-sur-Marne
  - Research Site, Colmar
  - Research Site, Creil
  - Research Site, Évreux
  - Research Site, Fleury-Mérogis
  - Research Site, Foix
  - Research Site, Le Kremlin-Bicêtre
  - Research Site, Maubeuge
  - Research Site, Meaux
  - Research Site, Mont-de-Marsan
  - Research Site, Montbonnot-Saint-Martin
  - Research Site, Nîmes
  - Research Site, Olivet
  - Research Site, Paris
  - Research Site, Quimper
  - Research Site, Saint-Maurice
  - Research Site, Saint-Michel
  - Research Site, Tournan-en-Brie
  - Research Site, Valenciennes
  - Research Site, Vandœuvre-lès-Nancy
  - Research Site, Vichy
- Germany (26):
  - Research Site, Ansbach
  - Research Site, Aschaffenburg
  - Research Site, Bad Münder am Deister
  - Research Site, Berlin
  - Research Site, Bischofswerda
  - Research Site, Dresden
  - Research Site, Duisburg
  - Research Site, Düsseldorf
  - Research Site, Erlangen
  - Research Site, Frankfurt
  - Research Site, Freiburg im Breisgau
  - Research Site, Greifswald
  - Research Site, Hannoversch Münden
  - Research Site, Ingolstadt
  - Research Site, Jena
  - Research Site, Kaufbeuren
  - Research Site, Lüdenscheid
  - Research Site, Marktheidenfeld
  - Research Site, München
  - Research Site, Pfarrkirchen
  - Research Site, Pirmasens
  - Research Site, Regensburg
  - Research Site, Rostock
  - Research Site, Saarbrücken
  - Research Site, Tangermünde
  - Research Site, Waldshut
- Greece (5):
  - Research Site, Alexandroupoli
  - Research Site, Athens
  - Research Site, Ioannina
  - Research Site, Thessaloniki
  - Research Site, Véroia
- Hungary (7):
  - Research Site, Budapest
  - Research Site, Győr
  - Research Site, Miskolc
  - Research Site, Nyíregyháza
  - Research Site, Szeged
  - Research Site, Székesfehérvár
  - Research Site, Veszprém
- Research Site, Reykjavik, Iceland
- Research Site, Galway, Ireland
- Italy (9):
  - Research Site, Bergamo, BG
  - Research Site, Treviglio, BG
  - Research Site, Cremona, CR
  - Research Site, Genova, GE
  - Research Site, Lodi, LO
  - Research Site, Milan, Mi
  - Research Site, Rozzano, MI
  - Research Site, Reggio Calabria, RC
  - Research Site, Busto Arsizio, VA
- Mexico (7):
  - Research Site, México, D.f.
  - Research Site, Acapulco de Juárez, Guerrero
  - Research Site, Guadalajara, Jalisco
  - Research Site, Cuernavaca, Morelos
  - Research Site, Monterrey, Nuevo León
  - Research Site, Distrito Federal
  - Research Site, San Luis Potosí City
- Netherlands (16):
  - Research Site, 's-Hertogenbosch
  - Research Site, Alkmaar
  - Research Site, Almelo
  - Research Site, Amersfoort
  - Research Site, Amsterdam
  - Research Site, Arnhem
  - Research Site, Deventer
  - Research Site, Dordrecht
  - Research Site, Emmen
  - Research Site, Groningen
  - Research Site, Leeuwarden
  - Research Site, Nieuwegein
  - Research Site, Rotterdam
  - Research Site, Sittard
  - Research Site, The Hague
  - Research Site, Tilburg
- Norway (10):
  - Research Site, Bergen
  - Research Site, Drammen
  - Research Site, Fredrikstad
  - Research Site, Lillehammer
  - Research Site, Lorenskog
  - Research Site, Oslo
  - Research Site, Skien
  - Research Site, Stavanger
  - Research Site, Trondheim
  - Research Site, Tønsberg
- Poland (9):
  - Research Site, Bialystok
  - Research Site, Gdansk
  - Research Site, Katowice
  - Research Site, Krakow
  - Research Site, Lublin
  - Research Site, Opole
  - Research Site, Płock
  - Research Site, Rybnik
  - Research Site, Włocławek
- South Korea (2):
  - Research Site, Seongnam-si, Korea
  - Research Site, Seoul, Korea
- Sweden (16):
  - Research Site, Eksjö
  - Research Site, Eskilstuna
  - Research Site, Falun
  - Research Site, Gävle
  - Research Site, Gothenburg
  - Research Site, Jönköping
  - Research Site, Karlstad
  - Research Site, Linköping
  - Research Site, Lund
  - Research Site, Mölndal
  - Research Site, Norrköping
  - Research Site, Örebro
  - Research Site, Skövde
  - Research Site, Stockholm
  - Research Site, Trollhättan
  - Research Site, Uppsala
- Switzerland (6):
  - Research Site, Aarau
  - Research Site, Bern
  - Research Site, Geneva
  - Research Site, Lausanne
  - Research Site, Sankt Gallen
  - Research Site, Zurich
- Turkey (Türkiye) (8):
  - Research Site, Istanbul, Altunizade
  - Research Site, Cebeci, Ankara
  - Research Site, Kampus, Antalya
  - Research Site, Antalya, Arapsuyu
  - Research Site, Ankara, Besevler
  - Research Site, Izmir, Bornova
  - Research Site, Bursa, Gorukle
  - Research Site, Istanbul, Haydarpasa
- United Kingdom (19):
  - Research Site, Antrim, Northern Ireland
  - Research Site, Belfast, Northern Ireland
  - Research Site, Newry, Northern Ireland
  - Research Site, Omagh, Northern Ireland
  - Research Site, Bradford
  - Research Site, Dumfries
  - Research Site, Dundee
  - Research Site, Glasgow
  - Research Site, Hull
  - Research Site, Kilmarnock
  - Research Site, Leeds
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Middlesbrough
  - Research Site, Newcastle
  - Research Site, Plymouth
  - Research Site, Rhyl
  - Research Site, Sheffield
  - Research Site, Surrey

REFERENCES:
- [Derived] Fellstrom BC, Jardine AG, Schmieder RE, Holdaas H, Bannister K, Beutler J, Chae DW, Chevaile A, Cobbe SM, Gronhagen-Riska C, De Lima JJ, Lins R, Mayer G, McMahon AW, Parving HH, Remuzzi G, Samuelsson O, Sonkodi S, Sci D, Suleymanlar G, Tsakiris D, Tesar V, Todorov V, Wiecek A, Wuthrich RP, Gottlow M, Johnsson E, Zannad F; AURORA Study Group. Rosuvastatin and cardiovascular events in patients undergoing hemodialysis. N Engl J Med. 2009 Apr 2;360(14):1395-407. doi: 10.1056/NEJMoa0810177. Epub 2009 Mar 30. PMID 19332456

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited patients were male or female with end-stage renal failure aged 50 to 80 years, who had received regular chronic haemodialysis treatment (including haemofiltration and hemodiafiltration ) for at least 3 months. They were recruited from 280 sites in 25 countries; recruitment started on 16 January 2003 and finished on 24 November 2004.
Pre-assignment Details: After a two week screening period, eligible patients were randomly assigned to either rosuvastatin treatment (10mg/day) or placebo with a 1:1 randomisation ratio. Follow-up was planned to continue until the accrual of 805 major cardiovascular events
Groups:
- Rosuvastatin 10mg: Rosuvastatin 10 mg oral tablets
Period: Overall Study
Arm/Group | Rosuvastatin 10mg | Placebo
Started | 1389 (Two patients were incorrectly randomised and not included in the analyses.) | 1384 (One patient was incorrectly randomised and not included in the analyses)
Completed | 1263 (Vital status was obtained for all randomised patients at the end of the study) | 1250 (Vital status was obtained for all randomised patients at the end of the study)
Not Completed | 126 | 134
Not completed — Withdrawal by Subject | 125 | 132
Not completed — Option selected by investigator | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rosuvastatin 10mg | Placebo | Total
Number analyzed (Participants) | 1389 | 1384 | 2773
Age Continuous [Mean (Standard Deviation); unit: Years] | 64.1 (8.6) | 64.3 (8.7) | 64.2 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 538 | 512 | 1050
  Male | 851 | 872 | 1723

OUTCOME MEASURES:

1. Primary Outcome: Number of Randomised Participants With a Major Cardiovascular Event (Non-fatal Stroke, Non-fatal Myocardial Infarction or Cardiovascular Death)
Time Frame: Events were reported continuously during the study. Duration of follow-up ranged from 1 day to 5.6 years
Measure: Number; unit: Participants
Arm/Group | Rosuvastatin 10mg | Placebo
Number analyzed (Participants) | 1389 | 1384
Participants | 396 | 408

2. Secondary Outcome: Number of Randomised Participants That Died From Any Cause.
Time Frame: Events were reported continuously during the study. Duration of follow-up ranged from 1 day to 5.6 years
Measure: Number; unit: Participants
Arm/Group | Rosuvastatin 10mg | Placebo
Number analyzed (Participants) | 1389 | 1384
Participants | 636 | 660

3. Secondary Outcome: Number of Randomised Participants With a Major Cardiovascular Event or That Died From Any Known Cause
Time Frame: Events were reported continuously during the study. Duration of follow-up ranged from 1 day to 5.6 years
Measure: Number; unit: Participants
Arm/Group | Rosuvastatin 10mg | Placebo
Number analyzed (Participants) | 1389 | 1384
Participants | 614 | 645

4. Secondary Outcome: Number of Randomised Participants That Died From Cardiovascular Cause
Time Frame: Events were reported continuously during the study. Duration of follow-up ranged from 1 day to 5.6 years
Measure: Number; unit: Participants
Arm/Group | Rosuvastatin 10mg | Placebo
Number analyzed (Participants) | 1389 | 1384
Participants | 324 | 324

5. Secondary Outcome: Number of Randomised Participants That Died From Non Cardiovascular Cause
Time Frame: Events were reported continuously during the study. Duration of follow-up ranged from 1 day to 5.6 years
Reporting Status: Not Posted
Measure: Number; unit: Participants

6. Secondary Outcome: Number of Randomised Participants With an Atherosclerotic Cardiac Event (Non-fatal Myocardial Infarction or Coronary Heart Disease (CHD) Death)
Time Frame: Events were reported continuously during the study. Duration of follow-up ranged from 1 day to 5.6 years
Measure: Number; unit: Participants
Arm/Group | Rosuvastatin 10mg | Placebo
Number analyzed (Participants) | 1389 | 1384
Participants | 258 | 256

7. Secondary Outcome: Number of Randomised Participants That Experienced a Procedure as a Result of Stenosis or Thrombosis of the Vascular Access (Arteriovenous (AV) Fistulas and Grafts Only) for Haemodialysis.
Time Frame: Events were reported continuously during the study. Duration of follow-up ranged from 1 day to 5.6 years
Measure: Number; unit: Participants
Arm/Group | Rosuvastatin 10mg | Placebo
Number analyzed (Participants) | 1389 | 1384
Participants | 390 | 360

8. Secondary Outcome: Number of Randomised Participants That Experienced a Coronary or Peripheral Revascularisation (Including Above Ankle Limb Amputations).
Time Frame: Events were reported continuously during the study. Duration of follow-up ranged from 1 day to 5.6 years
Measure: Number; unit: Participants
Arm/Group | Rosuvastatin 10mg | Placebo
Number analyzed (Participants) | 1389 | 1384
Participants | 148 | 152

ADVERSE EVENTS:
Description: The Participant flow chart shows the ITT Population (all correctly randomized patients) and is correct. The adverse event denominator represents the safety population, all randomized patients who received study drug. Six placebo patients never received treatment. This explains the apparent discrepancy.
Arm/Group | Rosuvastatin 10mg | Placebo
Serious Adverse Events (participants affected / at risk) | 1140 | 1159
Other Adverse Events (participants affected / at risk) | 620/1389 | 635/1378
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Rosuvastatin 10mg | Placebo
Convulsion (Nervous system disorders) | 6/1389 | 2/1378
Thrombocytopenia (Blood and lymphatic system disorders) | 1/1389 | 2/1378
Nephrogenic Anaemia (Blood and lymphatic system disorders) | 2/1389 | 1/1378
Coagulopathy (Blood and lymphatic system disorders) | 0/1389 | 1/1378
Haemolytic Anaemia (Blood and lymphatic system disorders) | 0/1389 | 1/1378
Haemorrhagic Diathesis (Blood and lymphatic system disorders) | 0/1389 | 1/1378
Pancytopenia (Blood and lymphatic system disorders) | 0/1389 | 1/1378
Splenic Infarction (Blood and lymphatic system disorders) | 0/1389 | 1/1378
Anaemia Megaloblastic (Blood and lymphatic system disorders) | 1/1389 | 0/1378
Lymphadenopathy Mediastinal (Blood and lymphatic system disorders) | 1/1389 | 0/1378
Polycythaemia (Blood and lymphatic system disorders) | 1/1389 | 0/1378
Myocardial Infarction (Cardiac disorders) | 53/1389 | 52/1378
Atrial Fibrillation (Cardiac disorders) | 39/1389 | 45/1378
Cardiac Failure (Cardiac disorders) | 30/1389 | 35/1378
Angina Pectoris (Cardiac disorders) | 21/1389 | 31/1378
Cardiac Arrest (Cardiac disorders) | 22/1389 | 26/1378
Acute Myocardial Infarction (Cardiac disorders) | 13/1389 | 10/1378
Cardiac Failure Congestive (Cardiac disorders) | 7/1389 | 12/1378
Bradycardia (Cardiac disorders) | 12/1389 | 5/1378
Angina Unstable (Cardiac disorders) | 9/1389 | 10/1378
Myocardial Ischaemia (Cardiac disorders) | 6/1389 | 10/1378
Atrioventricular Block Complete (Cardiac disorders) | 10/1389 | 6/1378
Coronary Artery Disease (Cardiac disorders) | 10/1389 | 7/1378
Arrhythmia (Cardiac disorders) | 8/1389 | 9/1378
Acute Coronary Syndrome (Cardiac disorders) | 9/1389 | 5/1378
Aortic Valve Stenosis (Cardiac disorders) | 8/1389 | 5/1378
Cardio-Respiratory Arrest (Cardiac disorders) | 6/1389 | 5/1378
Coronary Artery Stenosis (Cardiac disorders) | 6/1389 | 4/1378
Ventricular Tachycardia (Cardiac disorders) | 6/1389 | 3/1378
Cardiac Failure Acute (Cardiac disorders) | 5/1389 | 5/1378
Tachycardia (Cardiac disorders) | 1/1389 | 4/1378
Atrioventricular Block (Cardiac disorders) | 4/1389 | 1/1378
Ventricular Fibrillation (Cardiac disorders) | 4/1389 | 1/1378
Atrial Flutter (Cardiac disorders) | 3/1389 | 3/1378
Cardiac Asthma (Cardiac disorders) | 1/1389 | 3/1378
Cardiogenic Shock (Cardiac disorders) | 2/1389 | 3/1378
Hypertensive Cardiomyopathy (Cardiac disorders) | 0/1389 | 3/1378
Acute Left Ventricular Failure (Cardiac disorders) | 3/1389 | 0/1378
Pericarditis (Cardiac disorders) | 3/1389 | 0/1378
Sick Sinus Syndrome (Cardiac disorders) | 3/1389 | 0/1378
Supraventricular Tachycardia (Cardiac disorders) | 3/1389 | 1/1378
Cardiopulmonary Failure (Cardiac disorders) | 2/1389 | 2/1378
Congestive Cardiomyopathy (Cardiac disorders) | 2/1389 | 2/1378
Pericardial Effusion (Cardiac disorders) | 0/1389 | 2/1378
Atrioventricular Block Second Degree (Cardiac disorders) | 2/1389 | 0/1378
Cardiac Tamponade (Cardiac disorders) | 2/1389 | 0/1378
Palpitations (Cardiac disorders) | 2/1389 | 0/1378
Arrhythmia Supraventricular (Cardiac disorders) | 0/1389 | 1/1378
Bundle Branch Block Right (Cardiac disorders) | 0/1389 | 1/1378
Coronary Artery Insufficiency (Cardiac disorders) | 0/1389 | 1/1378
Ischaemic Cardiomyopathy (Cardiac disorders) | 0/1389 | 1/1378
Pericarditis Constrictive (Cardiac disorders) | 0/1389 | 1/1378
Prinzmetal Angina (Cardiac disorders) | 0/1389 | 1/1378
Right Ventricular Failure (Cardiac disorders) | 0/1389 | 1/1378
Silent Myocardial Infarction (Cardiac disorders) | 0/1389 | 1/1378
Sinus Arrhythmia (Cardiac disorders) | 0/1389 | 1/1378
Sinus Bradycardia (Cardiac disorders) | 0/1389 | 1/1378
Sinus Tachycardia (Cardiac disorders) | 0/1389 | 1/1378
Trifascicular Block (Cardiac disorders) | 0/1389 | 1/1378
Ventricular Extrasystoles (Cardiac disorders) | 1/1389 | 1/1378
Atrioventricular Block First Degree (Cardiac disorders) | 1/1389 | 0/1378
Cardiac Failure Chronic (Cardiac disorders) | 1/1389 | 0/1378
Cardiac Failure High Output (Cardiac disorders) | 1/1389 | 0/1378
Diastolic Dysfunction (Cardiac disorders) | 1/1389 | 0/1378
Hypertensive Heart Disease (Cardiac disorders) | 1/1389 | 0/1378
Nodal Rhythm (Cardiac disorders) | 1/1389 | 0/1378
Pericardial Haemorrhage (Cardiac disorders) | 1/1389 | 0/1378
Tachyarrhythmia (Cardiac disorders) | 1/1389 | 0/1378
Torsade De Pointes (Cardiac disorders) | 1/1389 | 0/1378
Ventricular Arrhythmia (Cardiac disorders) | 1/1389 | 0/1378
Atrial Septal Defect (Congenital, familial and genetic disorders) | 0/1389 | 1/1378
Gastrointestinal Angiodysplasia Haemorrhagic (Congenital, familial and genetic disorders) | 0/1389 | 1/1378
Gastrointestinal Angiodysplasia (Congenital, familial and genetic disorders) | 1/1389 | 0/1378
Polycystic Liver Disease (Congenital, familial and genetic disorders) | 1/1389 | 0/1378
Pyloric Stenosis (Congenital, familial and genetic disorders) | 1/1389 | 0/1378
Meniere's Disease (Ear and labyrinth disorders) | 0/1389 | 1/1378
Sudden Hearing Loss (Ear and labyrinth disorders) | 0/1389 | 1/1378
Tinnitus (Ear and labyrinth disorders) | 0/1389 | 1/1378
Vertigo (Ear and labyrinth disorders) | 1/1389 | 1/1378
Vertigo Positional (Ear and labyrinth disorders) | 1/1389 | 0/1378
Hyperparathyroidism (Endocrine disorders) | 18/1389 | 9/1378
Hyperparathyroidism Secondary (Endocrine disorders) | 7/1389 | 7/1378
Hyperparathyroidism Tertiary (Endocrine disorders) | 3/1389 | 1/1378
Hyperthyroidism (Endocrine disorders) | 0/1389 | 2/1378
Hypopituitarism (Endocrine disorders) | 1/1389 | 0/1378
Cataract (Eye disorders) | 16/1389 | 11/1378
Vitreous Haemorrhage (Eye disorders) | 3/1389 | 3/1378
Angle Closure Glaucoma (Eye disorders) | 2/1389 | 1/1378
Glaucoma (Eye disorders) | 2/1389 | 1/1378
Papilloedema (Eye disorders) | 1/1389 | 1/1378
Retinal Detachment (Eye disorders) | 0/1389 | 1/1378
Retinal Vein Occlusion (Eye disorders) | 0/1389 | 1/1378
Retinopathy (Eye disorders) | 0/1389 | 1/1378
Diabetic Retinopathy (Eye disorders) | 1/1389 | 0/1378
Diplopia (Eye disorders) | 1/1389 | 0/1378
Endophthalmitis (Eye disorders) | 1/1389 | 0/1378
Eye Haemorrhage (Eye disorders) | 1/1389 | 0/1378
Retinal Artery Occlusion (Eye disorders) | 1/1389 | 0/1378
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 25/1389 | 18/1378
Abdominal Pain (Gastrointestinal disorders) | 17/1389 | 12/1378
Diarrhoea (Gastrointestinal disorders) | 13/1389 | 9/1378
Gastritis (Gastrointestinal disorders) | 9/1389 | 4/1378
Peritonitis (Gastrointestinal disorders) | 9/1389 | 8/1378
Oesophagitis (Gastrointestinal disorders) | 2/1389 | 8/1378
Vomiting (Gastrointestinal disorders) | 7/1389 | 7/1378
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 2/1389 | 6/1378
Abdominal Pain Upper (Gastrointestinal disorders) | 5/1389 | 5/1378
Colitis Ischaemic (Gastrointestinal disorders) | 3/1389 | 5/1378
Duodenal Ulcer Haemorrhage (Gastrointestinal disorders) | 1/1389 | 5/1378
Gastric Ulcer Haemorrhage (Gastrointestinal disorders) | 5/1389 | 5/1378
Gastritis Erosive (Gastrointestinal disorders) | 1/1389 | 5/1378
Inguinal Hernia (Gastrointestinal disorders) | 1/1389 | 5/1378
Melaena (Gastrointestinal disorders) | 5/1389 | 5/1378
Gastric Ulcer (Gastrointestinal disorders) | 4/1389 | 4/1378
Haematemesis (Gastrointestinal disorders) | 4/1389 | 4/1378
Ileus (Gastrointestinal disorders) | 2/1389 | 4/1378
Colitis (Gastrointestinal disorders) | 4/1389 | 1/1378
Intestinal Ischaemia (Gastrointestinal disorders) | 4/1389 | 1/1378
Subileus (Gastrointestinal disorders) | 4/1389 | 0/1378
Colonic Polyp (Gastrointestinal disorders) | 3/1389 | 3/1378
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 3/1389 | 3/1378
Pancreatitis (Gastrointestinal disorders) | 2/1389 | 3/1378
Rectal Haemorrhage (Gastrointestinal disorders) | 3/1389 | 3/1378
Small Intestinal Obstruction (Gastrointestinal disorders) | 0/1389 | 3/1378
Constipation (Gastrointestinal disorders) | 3/1389 | 2/1378
Diverticulum Intestinal (Gastrointestinal disorders) | 3/1389 | 0/1378
Duodenal Ulcer (Gastrointestinal disorders) | 3/1389 | 2/1378
Intestinal Haemorrhage (Gastrointestinal disorders) | 3/1389 | 1/1378
Abdominal Symptom (Gastrointestinal disorders) | 0/1389 | 2/1378
Enteritis (Gastrointestinal disorders) | 0/1389 | 2/1378
Gastric Polyps (Gastrointestinal disorders) | 0/1389 | 2/1378
Intra-Abdominal Haemorrhage (Gastrointestinal disorders) | 2/1389 | 2/1378
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0/1389 | 2/1378
Sigmoiditis (Gastrointestinal disorders) | 0/1389 | 2/1378
Umbilical Hernia (Gastrointestinal disorders) | 1/1389 | 2/1378
Ascites (Gastrointestinal disorders) | 2/1389 | 1/1378
Intestinal Infarction (Gastrointestinal disorders) | 2/1389 | 1/1378
Intestinal Obstruction (Gastrointestinal disorders) | 2/1389 | 1/1378
Nausea (Gastrointestinal disorders) | 2/1389 | 1/1378
Peptic Ulcer (Gastrointestinal disorders) | 2/1389 | 0/1378
Colonic Pseudo-Obstruction (Gastrointestinal disorders) | 0/1389 | 1/1378
Crohn's Disease (Gastrointestinal disorders) | 0/1389 | 1/1378
Diverticulum (Gastrointestinal disorders) | 0/1389 | 1/1378
Dyspepsia (Gastrointestinal disorders) | 1/1389 | 1/1378
Enterocolitis (Gastrointestinal disorders) | 0/1389 | 1/1378
Enterocutaneous Fistula (Gastrointestinal disorders) | 0/1389 | 1/1378
Enterovesical Fistula (Gastrointestinal disorders) | 0/1389 | 1/1378
Faecaloma (Gastrointestinal disorders) | 1/1389 | 1/1378
Gastric Haemorrhage (Gastrointestinal disorders) | 1/1389 | 1/1378
Gastric Stenosis (Gastrointestinal disorders) | 0/1389 | 1/1378
Gastric Ulcer Perforation (Gastrointestinal disorders) | 0/1389 | 1/1378
Gastritis Haemorrhagic (Gastrointestinal disorders) | 1/1389 | 1/1378
Gastrointestinal Ischaemia (Gastrointestinal disorders) | 0/1389 | 1/1378
Gastrointestinal Perforation (Gastrointestinal disorders) | 1/1389 | 1/1378
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0/1389 | 1/1378
Haematochezia (Gastrointestinal disorders) | 1/1389 | 1/1378
Haemorrhoids (Gastrointestinal disorders) | 0/1389 | 1/1378
Ileitis (Gastrointestinal disorders) | 0/1389 | 1/1378
Impaired Gastric Emptying (Gastrointestinal disorders) | 1/1389 | 1/1378
Inguinal Hernia, Obstructive (Gastrointestinal disorders) | 0/1389 | 1/1378
Intestinal Angina (Gastrointestinal disorders) | 0/1389 | 1/1378
Intestinal Perforation (Gastrointestinal disorders) | 0/1389 | 1/1378
Intra-Abdominal Haematoma (Gastrointestinal disorders) | 0/1389 | 1/1378
Large Intestine Perforation (Gastrointestinal disorders) | 0/1389 | 1/1378
Mechanical Ileus (Gastrointestinal disorders) | 0/1389 | 1/1378
Mesenteric Artery Embolism (Gastrointestinal disorders) | 1/1389 | 1/1378
Mesenteric Vascular Insufficiency (Gastrointestinal disorders) | 0/1389 | 1/1378
Mouth Haemorrhage (Gastrointestinal disorders) | 0/1389 | 1/1378
Oesophagitis Haemorrhagic (Gastrointestinal disorders) | 0/1389 | 1/1378
Pancreatic Cyst (Gastrointestinal disorders) | 1/1389 | 1/1378
Periodontitis (Gastrointestinal disorders) | 1/1389 | 1/1378
Proctocolitis (Gastrointestinal disorders) | 0/1389 | 1/1378
Rectal Polyp (Gastrointestinal disorders) | 1/1389 | 1/1378
Sclerosing Encapsulating Peritonitis (Gastrointestinal disorders) | 0/1389 | 1/1378
Abdominal Hernia (Gastrointestinal disorders) | 1/1389 | 0/1378
Acute Abdomen (Gastrointestinal disorders) | 1/1389 | 0/1378
Anal Fistula (Gastrointestinal disorders) | 1/1389 | 0/1378
Dental Caries (Gastrointestinal disorders) | 1/1389 | 0/1378
Diarrhoea Haemorrhagic (Gastrointestinal disorders) | 1/1389 | 0/1378
Diverticular Perforation (Gastrointestinal disorders) | 1/1389 | 0/1378
Duodenitis (Gastrointestinal disorders) | 1/1389 | 0/1378
Food Poisoning (Gastrointestinal disorders) | 1/1389 | 0/1378
Gastroduodenitis (Gastrointestinal disorders) | 1/1389 | 0/1378
Gastrointestinal Motility Disorder (Gastrointestinal disorders) | 1/1389 | 0/1378
Gingival Bleeding (Gastrointestinal disorders) | 1/1389 | 0/1378
Ileus Paralytic (Gastrointestinal disorders) | 1/1389 | 0/1378
Intestinal Strangulation (Gastrointestinal disorders) | 1/1389 | 0/1378
Large Intestinal Haemorrhage (Gastrointestinal disorders) | 1/1389 | 0/1378
Mesenteric Artery Stenosis (Gastrointestinal disorders) | 1/1389 | 0/1378
Mesenteric Artery Thrombosis (Gastrointestinal disorders) | 1/1389 | 0/1378
Oesophageal Ulcer (Gastrointestinal disorders) | 1/1389 | 0/1378
Oesophageal Varices Haemorrhage (Gastrointestinal disorders) | 1/1389 | 0/1378
Pancreatitis Acute (Gastrointestinal disorders) | 1/1389 | 0/1378
Peritoneal Effusion (Gastrointestinal disorders) | 1/1389 | 0/1378
Reflux Oesophagitis (Gastrointestinal disorders) | 1/1389 | 0/1378
Retroperitoneal Effusion (Gastrointestinal disorders) | 1/1389 | 0/1378
Retroperitoneal Haematoma (Gastrointestinal disorders) | 1/1389 | 0/1378
Varices Oesophageal (Gastrointestinal disorders) | 1/1389 | 0/1378
Sudden Death (General disorders) | 33/1389 | 30/1378
Death (General disorders) | 30/1389 | 30/1378
Catheter Related Complication (General disorders) | 14/1389 | 17/1378
Pyrexia (General disorders) | 13/1389 | 15/1378
Catheter Thrombosis (General disorders) | 4/1389 | 10/1378
Malaise (General disorders) | 5/1389 | 10/1378
Sudden Cardiac Death (General disorders) | 8/1389 | 2/1378
Catheter Site Haemorrhage (General disorders) | 5/1389 | 7/1378
General Physical Health Deterioration (General disorders) | 4/1389 | 7/1378
Non-Cardiac Chest Pain (General disorders) | 6/1389 | 2/1378
Chest Pain (General disorders) | 3/1389 | 5/1378
Asthenia (General disorders) | 3/1389 | 3/1378
Cardiac Death (General disorders) | 2/1389 | 3/1378
Chills (General disorders) | 0/1389 | 3/1378
Discomfort (General disorders) | 2/1389 | 3/1378
Fatigue (General disorders) | 3/1389 | 3/1378
Inflammation (General disorders) | 1/1389 | 2/1378
Multi-Organ Failure (General disorders) | 1/1389 | 2/1378
Oedema Peripheral (General disorders) | 2/1389 | 2/1378
Wound Necrosis (General disorders) | 2/1389 | 2/1378
Gait Disturbance (General disorders) | 2/1389 | 0/1378
Catheter Site Haematoma (General disorders) | 0/1389 | 1/1378
Catheter Site Inflammation (General disorders) | 0/1389 | 1/1378
Haemorrhagic Cyst (General disorders) | 0/1389 | 1/1378
Hyperpyrexia (General disorders) | 1/1389 | 1/1378
Ulcer Haemorrhage (General disorders) | 0/1389 | 1/1378
Chest Discomfort (General disorders) | 1/1389 | 0/1378
Drug Interaction (General disorders) | 1/1389 | 0/1378
Hypothermia (General disorders) | 1/1389 | 0/1378
Influenza Like Illness (General disorders) | 1/1389 | 0/1378
Necrosis (General disorders) | 1/1389 | 0/1378
Pain (General disorders) | 1/1389 | 0/1378
Systemic Inflammatory Response Syndrome (General disorders) | 1/1389 | 0/1378
Cholelithiasis (Hepatobiliary disorders) | 9/1389 | 2/1378
Cholecystitis (Hepatobiliary disorders) | 5/1389 | 5/1378
Cholecystitis Acute (Hepatobiliary disorders) | 2/1389 | 2/1378
Biliary Dilatation (Hepatobiliary disorders) | 2/1389 | 0/1378
Cholangitis (Hepatobiliary disorders) | 2/1389 | 1/1378
Bile Duct Stone (Hepatobiliary disorders) | 1/1389 | 1/1378
Gallbladder Perforation (Hepatobiliary disorders) | 0/1389 | 1/1378
Hepatic Cyst (Hepatobiliary disorders) | 0/1389 | 1/1378
Hepatitis (Hepatobiliary disorders) | 1/1389 | 1/1378
Hepatitis Toxic (Hepatobiliary disorders) | 0/1389 | 1/1378
Jaundice (Hepatobiliary disorders) | 0/1389 | 1/1378
Bile Duct Obstruction (Hepatobiliary disorders) | 1/1389 | 0/1378
Biliary Colic (Hepatobiliary disorders) | 1/1389 | 0/1378
Cholecystitis Chronic (Hepatobiliary disorders) | 1/1389 | 0/1378
Hepatic Cirrhosis (Hepatobiliary disorders) | 1/1389 | 0/1378
Hepatic Function Abnormal (Hepatobiliary disorders) | 1/1389 | 0/1378
Hepatic Necrosis (Hepatobiliary disorders) | 1/1389 | 0/1378
Hyperbilirubinaemia (Hepatobiliary disorders) | 1/1389 | 0/1378
Portal Vein Occlusion (Hepatobiliary disorders) | 1/1389 | 0/1378
Anaphylactic Reaction (Immune system disorders) | 0/1389 | 2/1378
Amyloidosis (Immune system disorders) | 0/1389 | 1/1378
Kidney Transplant Rejection (Immune system disorders) | 0/1389 | 1/1378
Anaphylactic Shock (Immune system disorders) | 1/1389 | 0/1378
Pneumonia (Infections and infestations) | 92/1389 | 96/1378
Sepsis (Infections and infestations) | 65/1389 | 70/1378
Bronchitis (Infections and infestations) | 20/1389 | 22/1378
Bronchopneumonia (Infections and infestations) | 19/1389 | 18/1378
Gastroenteritis (Infections and infestations) | 19/1389 | 12/1378
Urinary Tract Infection (Infections and infestations) | 16/1389 | 10/1378
Catheter Related Infection (Infections and infestations) | 14/1389 | 15/1378
Arteriovenous Fistula Site Infection (Infections and infestations) | 15/1389 | 13/1378
Gangrene (Infections and infestations) | 10/1389 | 14/1378
Septic Shock (Infections and infestations) | 13/1389 | 9/1378
Cellulitis (Infections and infestations) | 11/1389 | 11/1378
Staphylococcal Sepsis (Infections and infestations) | 10/1389 | 11/1378
Respiratory Tract Infection (Infections and infestations) | 6/1389 | 10/1378
Arthritis Bacterial (Infections and infestations) | 3/1389 | 9/1378
Bacteraemia (Infections and infestations) | 9/1389 | 8/1378
Lobar Pneumonia (Infections and infestations) | 5/1389 | 8/1378
Localised Infection (Infections and infestations) | 8/1389 | 8/1378
Diverticulitis (Infections and infestations) | 5/1389 | 7/1378
Erysipelas (Infections and infestations) | 6/1389 | 7/1378
Viral Infection (Infections and infestations) | 7/1389 | 5/1378
Catheter Sepsis (Infections and infestations) | 4/1389 | 6/1378
Endocarditis (Infections and infestations) | 6/1389 | 6/1378
Infection (Infections and infestations) | 5/1389 | 6/1378
Lower Respiratory Tract Infection (Infections and infestations) | 6/1389 | 6/1378
Postoperative Wound Infection (Infections and infestations) | 6/1389 | 6/1378
Infected Skin Ulcer (Infections and infestations) | 6/1389 | 2/1378
Appendicitis (Infections and infestations) | 4/1389 | 5/1378
Arteriovenous Graft Site Infection (Infections and infestations) | 5/1389 | 5/1378
Clostridium Difficile Colitis (Infections and infestations) | 0/1389 | 5/1378
Osteomyelitis (Infections and infestations) | 5/1389 | 5/1378
Shunt Infection (Infections and infestations) | 3/1389 | 5/1378
Staphylococcal Infection (Infections and infestations) | 2/1389 | 5/1378
Central Line Infection (Infections and infestations) | 5/1389 | 4/1378
Wound Infection (Infections and infestations) | 5/1389 | 3/1378
Catheter Site Infection (Infections and infestations) | 3/1389 | 4/1378
Lung Infection (Infections and infestations) | 4/1389 | 4/1378
Graft Infection (Infections and infestations) | 4/1389 | 1/1378
Cystitis (Infections and infestations) | 0/1389 | 3/1378
Hepatitis C (Infections and infestations) | 0/1389 | 3/1378
Herpes Zoster (Infections and infestations) | 2/1389 | 3/1378
Intervertebral Discitis (Infections and infestations) | 1/1389 | 3/1378
Staphylococcal Bacteraemia (Infections and infestations) | 2/1389 | 3/1378
Arthritis Infective (Infections and infestations) | 3/1389 | 1/1378
Bacterial Infection (Infections and infestations) | 3/1389 | 0/1378
Device Related Infection (Infections and infestations) | 3/1389 | 1/1378
Gastroenteritis Viral (Infections and infestations) | 3/1389 | 0/1378
Post Procedural Infection (Infections and infestations) | 3/1389 | 1/1378
Postoperative Abscess (Infections and infestations) | 3/1389 | 0/1378
Renal Cyst Infection (Infections and infestations) | 3/1389 | 2/1378
Subcutaneous Abscess (Infections and infestations) | 3/1389 | 0/1378
Upper Respiratory Tract Infection (Infections and infestations) | 3/1389 | 0/1378
Abdominal Wall Abscess (Infections and infestations) | 0/1389 | 2/1378
Abscess Limb (Infections and infestations) | 1/1389 | 2/1378
Bacterial Sepsis (Infections and infestations) | 2/1389 | 2/1378
Diabetic Gangrene (Infections and infestations) | 2/1389 | 2/1378
Empyema (Infections and infestations) | 1/1389 | 2/1378
Endocarditis Bacterial (Infections and infestations) | 1/1389 | 2/1378
Enterococcal Sepsis (Infections and infestations) | 0/1389 | 2/1378
Hepatic Cyst Infection (Infections and infestations) | 2/1389 | 2/1378
Influenza (Infections and infestations) | 1/1389 | 2/1378
Meningitis (Infections and infestations) | 1/1389 | 2/1378
Nasopharyngitis (Infections and infestations) | 0/1389 | 2/1378
Pyelonephritis (Infections and infestations) | 2/1389 | 2/1378
Pyonephrosis (Infections and infestations) | 2/1389 | 2/1378
Skin Infection (Infections and infestations) | 2/1389 | 2/1378
Streptococcal Sepsis (Infections and infestations) | 0/1389 | 2/1378
Cytomegalovirus Infection (Infections and infestations) | 2/1389 | 1/1378
Pulmonary Tuberculosis (Infections and infestations) | 2/1389 | 1/1378
Tooth Infection (Infections and infestations) | 2/1389 | 1/1378
Abscess (Infections and infestations) | 0/1389 | 1/1378
Abscess Intestinal (Infections and infestations) | 0/1389 | 1/1378
Abscess Neck (Infections and infestations) | 0/1389 | 1/1378
Anal Abscess (Infections and infestations) | 0/1389 | 1/1378
Arteriosclerotic Gangrene (Infections and infestations) | 1/1389 | 1/1378
Bone Abscess (Infections and infestations) | 0/1389 | 1/1378
Bronchiectasis (Infections and infestations) | 0/1389 | 1/1378
Candida Sepsis (Infections and infestations) | 0/1389 | 1/1378
Escherichia Infection (Infections and infestations) | 1/1389 | 1/1378
Escherichia Sepsis (Infections and infestations) | 1/1389 | 1/1378
Febrile Infection (Infections and infestations) | 0/1389 | 1/1378
Fungal Sepsis (Infections and infestations) | 0/1389 | 1/1378
Gallbladder Abscess (Infections and infestations) | 0/1389 | 1/1378
Gallbladder Empyema (Infections and infestations) | 0/1389 | 1/1378
Groin Abscess (Infections and infestations) | 0/1389 | 1/1378
Haemophilus Infection (Infections and infestations) | 0/1389 | 1/1378
Helicobacter Gastritis (Infections and infestations) | 0/1389 | 1/1378
Hepatitis B (Infections and infestations) | 0/1389 | 1/1378
Hypopyon (Infections and infestations) | 0/1389 | 1/1378
Klebsiella Infection (Infections and infestations) | 0/1389 | 1/1378
Klebsiella Sepsis (Infections and infestations) | 1/1389 | 1/1378
Listeriosis (Infections and infestations) | 0/1389 | 1/1378
Liver Abscess (Infections and infestations) | 1/1389 | 1/1378
Mastoiditis (Infections and infestations) | 0/1389 | 1/1378
Myocarditis Septic (Infections and infestations) | 0/1389 | 1/1378
Oesophageal Candidiasis (Infections and infestations) | 1/1389 | 1/1378
Oral Fungal Infection (Infections and infestations) | 0/1389 | 1/1378
Orchitis (Infections and infestations) | 1/1389 | 1/1378
Pancreas Infection (Infections and infestations) | 0/1389 | 1/1378
Pelvic Abscess (Infections and infestations) | 0/1389 | 1/1378
Pelvic Infection (Infections and infestations) | 0/1389 | 1/1378
Penile Infection (Infections and infestations) | 0/1389 | 1/1378
Perinephric Abscess (Infections and infestations) | 1/1389 | 1/1378
Peritoneal Infection (Infections and infestations) | 0/1389 | 1/1378
Pneumonia Bacterial (Infections and infestations) | 1/1389 | 1/1378
Pneumonia Moraxella (Infections and infestations) | 0/1389 | 1/1378
Pneumonia Pneumococcal (Infections and infestations) | 0/1389 | 1/1378
Pseudomembranous Colitis (Infections and infestations) | 0/1389 | 1/1378
Pseudomonas Infection (Infections and infestations) | 0/1389 | 1/1378
Pyothorax (Infections and infestations) | 1/1389 | 1/1378
Rectal Abscess (Infections and infestations) | 0/1389 | 1/1378
Respiratory Tract Infection Viral (Infections and infestations) | 0/1389 | 1/1378
Salmonellosis (Infections and infestations) | 0/1389 | 1/1378
Scrotal Infection (Infections and infestations) | 0/1389 | 1/1378
Sepsis Syndrome (Infections and infestations) | 0/1389 | 1/1378
Streptococcal Bacteraemia (Infections and infestations) | 0/1389 | 1/1378
Streptococcal Infection (Infections and infestations) | 0/1389 | 1/1378
Tuberculosis (Infections and infestations) | 1/1389 | 1/1378
Urinary Tract Infection Staphylococcal (Infections and infestations) | 0/1389 | 1/1378
Urosepsis (Infections and infestations) | 1/1389 | 1/1378
Abdominal Infection (Infections and infestations) | 1/1389 | 0/1378
Abdominal Sepsis (Infections and infestations) | 1/1389 | 0/1378
Bronchitis Viral (Infections and infestations) | 1/1389 | 0/1378
Chronic Tonsillitis (Infections and infestations) | 1/1389 | 0/1378
Citrobacter Sepsis (Infections and infestations) | 1/1389 | 0/1378
Clostridial Infection (Infections and infestations) | 1/1389 | 0/1378
Clostridium Colitis (Infections and infestations) | 1/1389 | 0/1378
Diabetic Foot Infection (Infections and infestations) | 1/1389 | 0/1378
Diarrhoea Infectious (Infections and infestations) | 1/1389 | 0/1378
Endocarditis Staphylococcal (Infections and infestations) | 1/1389 | 0/1378
Enteritis Infectious (Infections and infestations) | 1/1389 | 0/1378
Escherichia Bacteraemia (Infections and infestations) | 1/1389 | 0/1378
Eye Infection (Infections and infestations) | 1/1389 | 0/1378
Fungal Infection (Infections and infestations) | 1/1389 | 0/1378
Furuncle (Infections and infestations) | 1/1389 | 0/1378
Herpes Simplex (Infections and infestations) | 1/1389 | 0/1378
Infective Exacerbation Of Chronic Obstructive Airways Disease (Infections and infestations) | 1/1389 | 0/1378
Infective Spondylitis (Infections and infestations) | 1/1389 | 0/1378
Lung Abscess (Infections and infestations) | 1/1389 | 0/1378
Lung Infection Pseudomonal (Infections and infestations) | 1/1389 | 0/1378
Meningitis Bacterial (Infections and infestations) | 1/1389 | 0/1378
Otitis Externa (Infections and infestations) | 1/1389 | 0/1378
Otitis Media (Infections and infestations) | 1/1389 | 0/1378
Peridiverticular Abscess (Infections and infestations) | 1/1389 | 0/1378
Perihepatic Abscess (Infections and infestations) | 1/1389 | 0/1378
Peritonitis Bacterial (Infections and infestations) | 1/1389 | 0/1378
Pneumococcal Sepsis (Infections and infestations) | 1/1389 | 0/1378
Pneumonia Klebsiella (Infections and infestations) | 1/1389 | 0/1378
Pseudomonal Sepsis (Infections and infestations) | 1/1389 | 0/1378
Pyelonephritis Acute (Infections and infestations) | 1/1389 | 0/1378
Respiratory Tract Infection Bacterial (Infections and infestations) | 1/1389 | 0/1378
Sinusitis (Infections and infestations) | 1/1389 | 0/1378
Toxoplasmosis (Infections and infestations) | 1/1389 | 0/1378
Tuberculous Pleurisy (Infections and infestations) | 1/1389 | 0/1378
Urinary Tract Infection Pseudomonal (Infections and infestations) | 1/1389 | 0/1378
Arteriovenous Fistula Site Complication (Injury, poisoning and procedural complications) | 54/1389 | 60/1378
Arteriovenous Fistula Thrombosis (Injury, poisoning and procedural complications) | 53/1389 | 45/1378
Vascular Access Complication (Injury, poisoning and procedural complications) | 30/1389 | 40/1378
Arteriovenous Fistula Site Haemorrhage (Injury, poisoning and procedural complications) | 20/1389 | 24/1378
Femur Fracture (Injury, poisoning and procedural complications) | 7/1389 | 19/1378
Arteriovenous Fistula Aneurysm (Injury, poisoning and procedural complications) | 13/1389 | 18/1378
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 13/1389 | 14/1378
Shunt Thrombosis (Injury, poisoning and procedural complications) | 12/1389 | 9/1378
Shunt Stenosis (Injury, poisoning and procedural complications) | 11/1389 | 4/1378
Vascular Graft Complication (Injury, poisoning and procedural complications) | 11/1389 | 8/1378
Graft Thrombosis (Injury, poisoning and procedural complications) | 4/1389 | 10/1378
Arteriovenous Graft Thrombosis (Injury, poisoning and procedural complications) | 10/1389 | 7/1378
Arteriovenous Fistula Occlusion (Injury, poisoning and procedural complications) | 4/1389 | 9/1378
Vascular Graft Occlusion (Injury, poisoning and procedural complications) | 4/1389 | 9/1378
Pelvic Fracture (Injury, poisoning and procedural complications) | 9/1389 | 7/1378
Haemodialysis-Induced Symptom (Injury, poisoning and procedural complications) | 3/1389 | 8/1378
Hip Fracture (Injury, poisoning and procedural complications) | 8/1389 | 4/1378
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 7/1389 | 3/1378
Procedural Hypotension (Injury, poisoning and procedural complications) | 7/1389 | 4/1378
Rib Fracture (Injury, poisoning and procedural complications) | 4/1389 | 6/1378
Fall (Injury, poisoning and procedural complications) | 6/1389 | 0/1378
Contusion (Injury, poisoning and procedural complications) | 1/1389 | 5/1378
Humerus Fracture (Injury, poisoning and procedural complications) | 4/1389 | 5/1378
Post Procedural Haematoma (Injury, poisoning and procedural complications) | 2/1389 | 5/1378
Shunt Occlusion (Injury, poisoning and procedural complications) | 2/1389 | 5/1378
Subdural Haematoma (Injury, poisoning and procedural complications) | 5/1389 | 3/1378
Wound (Injury, poisoning and procedural complications) | 5/1389 | 2/1378
Arteriovenous Fistula Site Haematoma (Injury, poisoning and procedural complications) | 4/1389 | 4/1378
Spinal Fracture (Injury, poisoning and procedural complications) | 4/1389 | 1/1378
Arteriovenous Graft Aneurysm (Injury, poisoning and procedural complications) | 1/1389 | 3/1378
Lower Limb Fracture (Injury, poisoning and procedural complications) | 1/1389 | 3/1378
Wrist Fracture (Injury, poisoning and procedural complications) | 0/1389 | 3/1378
Ankle Fracture (Injury, poisoning and procedural complications) | 3/1389 | 1/1378
Hand Fracture (Injury, poisoning and procedural complications) | 3/1389 | 1/1378
Post-Traumatic Pain (Injury, poisoning and procedural complications) | 3/1389 | 2/1378
Pubic Rami Fracture (Injury, poisoning and procedural complications) | 3/1389 | 2/1378
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 3/1389 | 2/1378
Tendon Rupture (Injury, poisoning and procedural complications) | 3/1389 | 1/1378
Arteriovenous Graft Site Haemorrhage (Injury, poisoning and procedural complications) | 0/1389 | 2/1378
Complications Of Transplanted Kidney (Injury, poisoning and procedural complications) | 0/1389 | 2/1378
Foot Fracture (Injury, poisoning and procedural complications) | 1/1389 | 2/1378
Head Injury (Injury, poisoning and procedural complications) | 2/1389 | 2/1378
Incisional Hernia (Injury, poisoning and procedural complications) | 0/1389 | 2/1378
Joint Dislocation (Injury, poisoning and procedural complications) | 1/1389 | 2/1378
Procedural Pain (Injury, poisoning and procedural complications) | 2/1389 | 2/1378
Shunt Malfunction (Injury, poisoning and procedural complications) | 2/1389 | 2/1378
Therapeutic Agent Toxicity (Injury, poisoning and procedural complications) | 2/1389 | 2/1378
Thoracic Vertebral Fracture (Injury, poisoning and procedural complications) | 0/1389 | 2/1378
Tibia Fracture (Injury, poisoning and procedural complications) | 2/1389 | 2/1378
Traumatic Haematoma (Injury, poisoning and procedural complications) | 0/1389 | 2/1378
Upper Limb Fracture (Injury, poisoning and procedural complications) | 1/1389 | 2/1378
Vascular Procedure Complication (Injury, poisoning and procedural complications) | 1/1389 | 2/1378
Vascular Pseudoaneurysm (Injury, poisoning and procedural complications) | 1/1389 | 2/1378
Accidental Overdose (Injury, poisoning and procedural complications) | 2/1389 | 0/1378
Arteriovenous Graft Site Haematoma (Injury, poisoning and procedural complications) | 2/1389 | 1/1378
Concussion (Injury, poisoning and procedural complications) | 2/1389 | 0/1378
Dialysis Device Complication (Injury, poisoning and procedural complications) | 2/1389 | 1/1378
Injury (Injury, poisoning and procedural complications) | 2/1389 | 1/1378
Postoperative Wound Complication (Injury, poisoning and procedural complications) | 2/1389 | 1/1378
Radius Fracture (Injury, poisoning and procedural complications) | 2/1389 | 1/1378
Road Traffic Accident (Injury, poisoning and procedural complications) | 2/1389 | 1/1378
Acetabulum Fracture (Injury, poisoning and procedural complications) | 1/1389 | 1/1378
Alcohol Poisoning (Injury, poisoning and procedural complications) | 0/1389 | 1/1378
Cerebral Haemorrhage Traumatic (Injury, poisoning and procedural complications) | 0/1389 | 1/1378
Cervical Vertebral Fracture (Injury, poisoning and procedural complications) | 0/1389 | 1/1378
Chest Injury (Injury, poisoning and procedural complications) | 0/1389 | 1/1378
Clavicle Fracture (Injury, poisoning and procedural complications) | 0/1389 | 1/1378
Extrusion Of Device (Injury, poisoning and procedural complications) | 0/1389 | 1/1378
Foreign Body Trauma (Injury, poisoning and procedural complications) | 0/1389 | 1/1378
Graft Complication (Injury, poisoning and procedural complications) | 1/1389 | 1/1378
Graft Haemorrhage (Injury, poisoning and procedural complications) | 0/1389 | 1/1378
Heat Illness (Injury, poisoning and procedural complications) | 0/1389 | 1/1378
Joint Injury (Injury, poisoning and procedural complications) | 1/1389 | 1/1378
Limb Injury (Injury, poisoning and procedural complications) | 1/1389 | 1/1378
Medical Device Complication (Injury, poisoning and procedural complications) | 1/1389 | 1/1378
Medical Device Pain (Injury, poisoning and procedural complications) | 0/1389 | 1/1378
Multiple Fractures (Injury, poisoning and procedural complications) | 0/1389 | 1/1378
Multiple Injuries (Injury, poisoning and procedural complications) | 1/1389 | 1/1378
Muscle Strain (Injury, poisoning and procedural complications) | 0/1389 | 1/1378
Narcotic Intoxication (Injury, poisoning and procedural complications) | 0/1389 | 1/1378
Overdose (Injury, poisoning and procedural complications) | 1/1389 | 1/1378
Patella Fracture (Injury, poisoning and procedural complications) | 0/1389 | 1/1378
Periorbital Haematoma (Injury, poisoning and procedural complications) | 0/1389 | 1/1378
Perirenal Haematoma (Injury, poisoning and procedural complications) | 0/1389 | 1/1378
Post Procedural Fistula (Injury, poisoning and procedural complications) | 0/1389 | 1/1378
Shunt Aneurysm (Injury, poisoning and procedural complications) | 0/1389 | 1/1378
Skeletal Injury (Injury, poisoning and procedural complications) | 0/1389 | 1/1378
Skin Laceration (Injury, poisoning and procedural complications) | 0/1389 | 1/1378
Sternal Fracture (Injury, poisoning and procedural complications) | 0/1389 | 1/1378
Thermal Burn (Injury, poisoning and procedural complications) | 1/1389 | 1/1378
Wound Dehiscence (Injury, poisoning and procedural complications) | 0/1389 | 1/1378
Anaemia Postoperative (Injury, poisoning and procedural complications) | 1/1389 | 0/1378
Arterial Injury (Injury, poisoning and procedural complications) | 1/1389 | 0/1378
Cardiac Pacemaker Malfunction (Injury, poisoning and procedural complications) | 1/1389 | 0/1378
Cardiac Procedure Complication (Injury, poisoning and procedural complications) | 1/1389 | 0/1378
Collapse Of Lung (Injury, poisoning and procedural complications) | 1/1389 | 0/1378
Comminuted Fracture (Injury, poisoning and procedural complications) | 1/1389 | 0/1378
Dialysis Disequilibrium Syndrome (Injury, poisoning and procedural complications) | 1/1389 | 0/1378
Dislocation Of Joint Prosthesis (Injury, poisoning and procedural complications) | 1/1389 | 0/1378
Dislocation Of Vertebra (Injury, poisoning and procedural complications) | 1/1389 | 0/1378
Drug Toxicity (Injury, poisoning and procedural complications) | 1/1389 | 0/1378
Facial Bones Fracture (Injury, poisoning and procedural complications) | 1/1389 | 0/1378
Fractured Sacrum (Injury, poisoning and procedural complications) | 1/1389 | 0/1378
Haemolytic Transfusion Reaction (Injury, poisoning and procedural complications) | 1/1389 | 0/1378
Ilium Fracture (Injury, poisoning and procedural complications) | 1/1389 | 0/1378
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 1/1389 | 0/1378
Operative Haemorrhage (Injury, poisoning and procedural complications) | 1/1389 | 0/1378
Pacemaker Complication (Injury, poisoning and procedural complications) | 1/1389 | 0/1378
Peripheral Nerve Injury (Injury, poisoning and procedural complications) | 1/1389 | 0/1378
Procedural Vomiting (Injury, poisoning and procedural complications) | 1/1389 | 0/1378
Skull Fracture (Injury, poisoning and procedural complications) | 1/1389 | 0/1378
Stent-Graft Endoleak (Injury, poisoning and procedural complications) | 1/1389 | 0/1378
Subdural Haemorrhage (Injury, poisoning and procedural complications) | 1/1389 | 0/1378
Suture Related Complication (Injury, poisoning and procedural complications) | 1/1389 | 0/1378
Transfusion Reaction (Injury, poisoning and procedural complications) | 1/1389 | 0/1378
Traumatic Brain Injury (Injury, poisoning and procedural complications) | 1/1389 | 0/1378
Traumatic Intracranial Haemorrhage (Injury, poisoning and procedural complications) | 1/1389 | 0/1378
Vascular Injury (Injury, poisoning and procedural complications) | 1/1389 | 0/1378
Venous Injury (Injury, poisoning and procedural complications) | 1/1389 | 0/1378
Weight Decreased (Injury, poisoning and procedural complications) | 1/1389 | 4/1378
International Normalised Ratio Increased (Injury, poisoning and procedural complications) | 0/1389 | 2/1378
Blood Calcium Decreased (Injury, poisoning and procedural complications) | 2/1389 | 0/1378
Blood Pressure Increased (Injury, poisoning and procedural complications) | 2/1389 | 0/1378
Blood Glucose Increased (Injury, poisoning and procedural complications) | 0/1389 | 1/1378
C-Reactive Protein Increased (Injury, poisoning and procedural complications) | 1/1389 | 1/1378
Electrocardiogram Q Wave Abnormal (Injury, poisoning and procedural complications) | 0/1389 | 1/1378
Electrocardiogram T Wave Inversion (Injury, poisoning and procedural complications) | 0/1389 | 1/1378
Occult Blood Positive (Injury, poisoning and procedural complications) | 0/1389 | 1/1378
Urine Cytology Abnormal (Injury, poisoning and procedural complications) | 0/1389 | 1/1378
Alanine Aminotransferase Increased (Injury, poisoning and procedural complications) | 1/1389 | 0/1378
Blood Creatinine Increased (Injury, poisoning and procedural complications) | 1/1389 | 0/1378
Blood Culture Positive (Injury, poisoning and procedural complications) | 1/1389 | 0/1378
Blood Potassium Increased (Injury, poisoning and procedural complications) | 1/1389 | 0/1378
Electrocardiogram T Wave Amplitude Increased (Injury, poisoning and procedural complications) | 1/1389 | 0/1378
Haemoglobin Decreased (Injury, poisoning and procedural complications) | 1/1389 | 0/1378
Liver Function Test Abnormal (Injury, poisoning and procedural complications) | 1/1389 | 0/1378
Hyperkalaemia (Metabolism and nutrition disorders) | 7/1389 | 13/1378
Diabetic Foot (Metabolism and nutrition disorders) | 3/1389 | 12/1378
Fluid Overload (Metabolism and nutrition disorders) | 7/1389 | 10/1378
Hypoglycaemia (Metabolism and nutrition disorders) | 7/1389 | 8/1378
Fluid Retention (Metabolism and nutrition disorders) | 8/1389 | 6/1378
Dehydration (Metabolism and nutrition disorders) | 4/1389 | 1/1378
Calciphylaxis (Metabolism and nutrition disorders) | 3/1389 | 3/1378
Malnutrition (Metabolism and nutrition disorders) | 2/1389 | 3/1378
Diabetes Mellitus (Metabolism and nutrition disorders) | 3/1389 | 2/1378
Hyperglycaemia (Metabolism and nutrition disorders) | 3/1389 | 0/1378
Cachexia (Metabolism and nutrition disorders) | 2/1389 | 2/1378
Hyperphosphataemia (Metabolism and nutrition disorders) | 1/1389 | 2/1378
Hypokalaemia (Metabolism and nutrition disorders) | 1/1389 | 2/1378
Hypervolaemia (Metabolism and nutrition disorders) | 2/1389 | 0/1378
Metabolic Acidosis (Metabolism and nutrition disorders) | 2/1389 | 1/1378
Anorexia (Metabolism and nutrition disorders) | 1/1389 | 1/1378
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 1/1389 | 1/1378
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 0/1389 | 1/1378
Gout (Metabolism and nutrition disorders) | 1/1389 | 1/1378
Hypocalcaemia (Metabolism and nutrition disorders) | 0/1389 | 1/1378
Hypovolaemia (Metabolism and nutrition disorders) | 0/1389 | 1/1378
Hypercalcaemia (Metabolism and nutrition disorders) | 1/1389 | 0/1378
Metabolic Disorder (Metabolism and nutrition disorders) | 1/1389 | 0/1378
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 8/1389 | 5/1378
Arthralgia (Musculoskeletal and connective tissue disorders) | 5/1389 | 7/1378
Arthritis (Musculoskeletal and connective tissue disorders) | 1/1389 | 7/1378
Back Pain (Musculoskeletal and connective tissue disorders) | 7/1389 | 7/1378
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 2/1389 | 4/1378
Neck Pain (Musculoskeletal and connective tissue disorders) | 4/1389 | 0/1378
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 4/1389 | 3/1378
Muscle Haemorrhage (Musculoskeletal and connective tissue disorders) | 1/1389 | 3/1378
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1/1389 | 3/1378
Osteitis (Musculoskeletal and connective tissue disorders) | 2/1389 | 3/1378
Bursitis (Musculoskeletal and connective tissue disorders) | 3/1389 | 1/1378
Spinal Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3/1389 | 0/1378
Bone Pain (Musculoskeletal and connective tissue disorders) | 1/1389 | 2/1378
Chondrocalcinosis Pyrophosphate (Musculoskeletal and connective tissue disorders) | 0/1389 | 2/1378
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 2/1389 | 0/1378
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 2/1389 | 1/1378
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0/1389 | 1/1378
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0/1389 | 1/1378
Myalgia (Musculoskeletal and connective tissue disorders) | 1/1389 | 1/1378
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0/1389 | 1/1378
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0/1389 | 1/1378
Polymyalgia Rheumatica (Musculoskeletal and connective tissue disorders) | 0/1389 | 1/1378
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0/1389 | 1/1378
Soft Tissue Haemorrhage (Musculoskeletal and connective tissue disorders) | 0/1389 | 1/1378
Synovial Cyst (Musculoskeletal and connective tissue disorders) | 0/1389 | 1/1378
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0/1389 | 1/1378
Trigger Finger (Musculoskeletal and connective tissue disorders) | 0/1389 | 1/1378
Bone Cyst (Musculoskeletal and connective tissue disorders) | 1/1389 | 0/1378
Dupuytren's Contracture (Musculoskeletal and connective tissue disorders) | 1/1389 | 0/1378
Intervertebral Disc Space Narrowing (Musculoskeletal and connective tissue disorders) | 1/1389 | 0/1378
Joint Swelling (Musculoskeletal and connective tissue disorders) | 1/1389 | 0/1378
Monarthritis (Musculoskeletal and connective tissue disorders) | 1/1389 | 0/1378
Nodal Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1/1389 | 0/1378
Osteitis Deformans (Musculoskeletal and connective tissue disorders) | 1/1389 | 0/1378
Psoriatic Arthropathy (Musculoskeletal and connective tissue disorders) | 1/1389 | 0/1378
Synovitis (Musculoskeletal and connective tissue disorders) | 1/1389 | 0/1378
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3/1389 | 7/1378
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/1389 | 4/1378
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/1389 | 4/1378
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4/1389 | 4/1378
Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/1389 | 4/1378
Metastases To Liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4/1389 | 1/1378
Parathyroid Tumour Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4/1389 | 0/1378
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3/1389 | 1/1378
Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3/1389 | 0/1378
Metastases To Lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3/1389 | 0/1378
Oesophageal Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/1389 | 2/1378
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/1389 | 2/1378
Rectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/1389 | 2/1378
Skin Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/1389 | 2/1378
Squamous Cell Carcinoma Of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/1389 | 2/1378
Hepatic Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/1389 | 0/1378
Lip Neoplasm Malignant Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/1389 | 0/1378
Lung Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/1389 | 1/1378
Rectosigmoid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/1389 | 0/1378
Renal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/1389 | 1/1378
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/1389 | 1/1378
Bile Duct Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/1389 | 1/1378
Bladder Transitional Cell Carcinoma Stage Iii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/1389 | 1/1378
Cervix Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/1389 | 1/1378
Colon Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/1389 | 1/1378
Colon Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/1389 | 1/1378
Epiglottic Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/1389 | 1/1378
Gallbladder Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/1389 | 1/1378
Gastrointestinal Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/1389 | 1/1378
Laryngeal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/1389 | 1/1378
Laryngeal Cancer Stage Iii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/1389 | 1/1378
Leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/1389 | 1/1378
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/1389 | 1/1378
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/1389 | 1/1378
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/1389 | 1/1378
Metastatic Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/1389 | 1/1378
Metastatic Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/1389 | 1/1378
Metastatic Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/1389 | 1/1378
Non-Hodgkin's Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/1389 | 1/1378
Prostate Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/1389 | 1/1378
Prostatic Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/1389 | 1/1378
Renal Oncocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/1389 | 1/1378
Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/1389 | 1/1378
Uterine Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/1389 | 1/1378
Benign Breast Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/1389 | 0/1378
Benign Lung Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/1389 | 0/1378
Benign Neoplasm Of Testis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/1389 | 0/1378
Benign Small Intestinal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/1389 | 0/1378
Bladder Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/1389 | 0/1378
Bone Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/1389 | 0/1378
Brain Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/1389 | 0/1378
Breast Cancer Female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/1389 | 0/1378
Carcinoid Tumour Of The Stomach (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/1389 | 0/1378
Choroid Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/1389 | 0/1378
Colon Cancer Stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/1389 | 0/1378
Follicle Centre Lymphoma, Follicular Grade I, Ii, Iii Stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/1389 | 0/1378
Gastrointestinal Tract Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/1389 | 0/1378
Liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/1389 | 0/1378
Lung Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/1389 | 0/1378
Lung Squamous Cell Carcinoma Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/1389 | 0/1378
Lymphocytic Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/1389 | 0/1378
Metastases To Central Nervous System (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/1389 | 0/1378
Metastatic Carcinoma Of The Bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/1389 | 0/1378
Metastatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/1389 | 0/1378
Multiple Myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/1389 | 0/1378
Non-Small Cell Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/1389 | 0/1378
Ovarian Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/1389 | 0/1378
Pancreatic Carcinoma Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/1389 | 0/1378
Rectal Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/1389 | 0/1378
Rectal Cancer Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/1389 | 0/1378
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/1389 | 0/1378
Tongue Neoplasm Malignant Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/1389 | 0/1378
Cerebrovascular Accident (Nervous system disorders) | 30/1389 | 29/1378
Carpal Tunnel Syndrome (Nervous system disorders) | 10/1389 | 10/1378
Syncope (Nervous system disorders) | 10/1389 | 7/1378
Haemorrhagic Stroke (Nervous system disorders) | 9/1389 | 1/1378
Cerebral Haemorrhage (Nervous system disorders) | 6/1389 | 8/1378
Ischaemic Stroke (Nervous system disorders) | 6/1389 | 8/1378
Cerebral Infarction (Nervous system disorders) | 2/1389 | 5/1378
Carotid Artery Stenosis (Nervous system disorders) | 4/1389 | 0/1378
Epilepsy (Nervous system disorders) | 2/1389 | 3/1378
Subarachnoid Haemorrhage (Nervous system disorders) | 3/1389 | 3/1378
Headache (Nervous system disorders) | 3/1389 | 1/1378
Dizziness (Nervous system disorders) | 1/1389 | 2/1378
Dysarthria (Nervous system disorders) | 2/1389 | 2/1378
Haemorrhage Intracranial (Nervous system disorders) | 2/1389 | 2/1378
Hypoglycaemic Coma (Nervous system disorders) | 0/1389 | 2/1378
Loss Of Consciousness (Nervous system disorders) | 1/1389 | 2/1378
Sciatica (Nervous system disorders) | 2/1389 | 2/1378
Somnolence (Nervous system disorders) | 1/1389 | 2/1378
Vertebrobasilar Insufficiency (Nervous system disorders) | 0/1389 | 2/1378
Carotid Arteriosclerosis (Nervous system disorders) | 2/1389 | 0/1378
Cerebellar Haemorrhage (Nervous system disorders) | 2/1389 | 1/1378
Coma (Nervous system disorders) | 2/1389 | 1/1378
Dementia (Nervous system disorders) | 2/1389 | 0/1378
Depressed Level Of Consciousness (Nervous system disorders) | 2/1389 | 0/1378
Grand Mal Convulsion (Nervous system disorders) | 2/1389 | 1/1378
Hypertensive Encephalopathy (Nervous system disorders) | 2/1389 | 1/1378
Uraemic Encephalopathy (Nervous system disorders) | 2/1389 | 0/1378
Balance Disorder (Nervous system disorders) | 0/1389 | 1/1378
Brain Oedema (Nervous system disorders) | 0/1389 | 1/1378
Cerebral Arteriosclerosis (Nervous system disorders) | 0/1389 | 1/1378
Cerebral Artery Thrombosis (Nervous system disorders) | 0/1389 | 1/1378
Cerebral Ischaemia (Nervous system disorders) | 1/1389 | 1/1378
Cerebrovascular Disorder (Nervous system disorders) | 0/1389 | 1/1378
Cervical Cord Compression (Nervous system disorders) | 0/1389 | 1/1378
Cognitive Disorder (Nervous system disorders) | 0/1389 | 1/1378
Coma Hepatic (Nervous system disorders) | 0/1389 | 1/1378
Coma Uraemic (Nervous system disorders) | 0/1389 | 1/1378
Demyelination (Nervous system disorders) | 0/1389 | 1/1378
Diabetic Neuropathy (Nervous system disorders) | 0/1389 | 1/1378
Encephalopathy (Nervous system disorders) | 1/1389 | 1/1378
Hemiplegia (Nervous system disorders) | 0/1389 | 1/1378
Lacunar Infarction (Nervous system disorders) | 0/1389 | 1/1378
Memory Impairment (Nervous system disorders) | 0/1389 | 1/1378
Nervous System Disorder (Nervous system disorders) | 1/1389 | 1/1378
Neuralgia (Nervous system disorders) | 1/1389 | 1/1378
Neurodegenerative Disorder (Nervous system disorders) | 0/1389 | 1/1378
Peripheral Motor Neuropathy (Nervous system disorders) | 0/1389 | 1/1378
Spondylitic Myelopathy (Nervous system disorders) | 0/1389 | 1/1378
Status Epilepticus (Nervous system disorders) | 0/1389 | 1/1378
Stupor (Nervous system disorders) | 1/1389 | 1/1378
Altered State Of Consciousness (Nervous system disorders) | 1/1389 | 0/1378
Amnesia (Nervous system disorders) | 1/1389 | 0/1378
Anoxic Encephalopathy (Nervous system disorders) | 1/1389 | 0/1378
Arachnoid Cyst (Nervous system disorders) | 1/1389 | 0/1378
Brain Compression (Nervous system disorders) | 1/1389 | 0/1378
Cerebral Disorder (Nervous system disorders) | 1/1389 | 0/1378
Diabetic Autonomic Neuropathy (Nervous system disorders) | 1/1389 | 0/1378
Guillain-Barre Syndrome (Nervous system disorders) | 1/1389 | 0/1378
Hemiparesis (Nervous system disorders) | 1/1389 | 0/1378
Hydrocephalus (Nervous system disorders) | 1/1389 | 0/1378
Hypoaesthesia (Nervous system disorders) | 1/1389 | 0/1378
Intercostal Neuralgia (Nervous system disorders) | 1/1389 | 0/1378
Intracranial Aneurysm (Nervous system disorders) | 1/1389 | 0/1378
Intracranial Haematoma (Nervous system disorders) | 1/1389 | 0/1378
Intraventricular Haemorrhage (Nervous system disorders) | 1/1389 | 0/1378
Metabolic Encephalopathy (Nervous system disorders) | 1/1389 | 0/1378
Monoparesis (Nervous system disorders) | 1/1389 | 0/1378
Neuropathy Peripheral (Nervous system disorders) | 1/1389 | 0/1378
Parkinson's Disease (Nervous system disorders) | 1/1389 | 0/1378
Presenile Dementia (Nervous system disorders) | 1/1389 | 0/1378
Quadriparesis (Nervous system disorders) | 1/1389 | 0/1378
Restless Legs Syndrome (Nervous system disorders) | 1/1389 | 0/1378
Simple Partial Seizures (Nervous system disorders) | 1/1389 | 0/1378
Vascular Dementia (Nervous system disorders) | 1/1389 | 0/1378
Vascular Encephalopathy (Nervous system disorders) | 1/1389 | 0/1378
Confusional State (Psychiatric disorders) | 6/1389 | 10/1378
Delirium (Psychiatric disorders) | 2/1389 | 2/1378
Sleep Disorder (Psychiatric disorders) | 2/1389 | 0/1378
Alcohol Abuse (Psychiatric disorders) | 0/1389 | 1/1378
Anxiety (Psychiatric disorders) | 1/1389 | 1/1378
Completed Suicide (Psychiatric disorders) | 0/1389 | 1/1378
Depression (Psychiatric disorders) | 0/1389 | 1/1378
Disorientation (Psychiatric disorders) | 1/1389 | 1/1378
Impaired Self-Care (Psychiatric disorders) | 0/1389 | 1/1378
Psychotic Disorder (Psychiatric disorders) | 1/1389 | 1/1378
Delusional Disorder, Persecutory Type (Psychiatric disorders) | 1/1389 | 0/1378
Insomnia (Psychiatric disorders) | 1/1389 | 0/1378
Mental Disorder (Psychiatric disorders) | 1/1389 | 0/1378
Psychotic Disorder Due To A General Medical Condition (Psychiatric disorders) | 1/1389 | 0/1378
Renal Failure Chronic (Renal and urinary disorders) | 8/1389 | 9/1378
Haematuria (Renal and urinary disorders) | 5/1389 | 8/1378
Azotaemia (Renal and urinary disorders) | 3/1389 | 4/1378
Renal Haemorrhage (Renal and urinary disorders) | 3/1389 | 1/1378
Renal Colic (Renal and urinary disorders) | 0/1389 | 2/1378
Renal Failure (Renal and urinary disorders) | 2/1389 | 2/1378
Calculus Bladder (Renal and urinary disorders) | 2/1389 | 0/1378
Renal Cyst (Renal and urinary disorders) | 2/1389 | 1/1378
Dysuria (Renal and urinary disorders) | 0/1389 | 1/1378
Extravasation Of Urine (Renal and urinary disorders) | 0/1389 | 1/1378
Hypertonic Bladder (Renal and urinary disorders) | 1/1389 | 1/1378
Pyuria (Renal and urinary disorders) | 0/1389 | 1/1378
Renal Artery Stenosis (Renal and urinary disorders) | 0/1389 | 1/1378
Ureteric Obstruction (Renal and urinary disorders) | 0/1389 | 1/1378
Urinary Retention (Renal and urinary disorders) | 0/1389 | 1/1378
Calculus Urethral (Renal and urinary disorders) | 1/1389 | 0/1378
Cystitis Haemorrhagic (Renal and urinary disorders) | 1/1389 | 0/1378
Hydronephrosis (Renal and urinary disorders) | 1/1389 | 0/1378
Nephrolithiasis (Renal and urinary disorders) | 1/1389 | 0/1378
Renal Cyst Ruptured (Renal and urinary disorders) | 1/1389 | 0/1378
Urethral Stenosis (Renal and urinary disorders) | 1/1389 | 0/1378
Urinary Bladder Haemorrhage (Renal and urinary disorders) | 1/1389 | 0/1378
Metrorrhagia (Reproductive system and breast disorders) | 0/1389 | 2/1378
Prostatism (Reproductive system and breast disorders) | 2/1389 | 0/1378
Prostatomegaly (Reproductive system and breast disorders) | 2/1389 | 0/1378
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 1/1389 | 1/1378
Endometrial Hypertrophy (Reproductive system and breast disorders) | 0/1389 | 1/1378
Menorrhagia (Reproductive system and breast disorders) | 0/1389 | 1/1378
Ovarian Cyst (Reproductive system and breast disorders) | 1/1389 | 1/1378
Pelvic Pain (Reproductive system and breast disorders) | 0/1389 | 1/1378
Prostatitis (Reproductive system and breast disorders) | 1/1389 | 1/1378
Uterine Prolapse (Reproductive system and breast disorders) | 0/1389 | 1/1378
Balanitis (Reproductive system and breast disorders) | 1/1389 | 0/1378
Dysfunctional Uterine Bleeding (Reproductive system and breast disorders) | 1/1389 | 0/1378
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 13/1389 | 25/1378
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 19/1389 | 22/1378
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 6/1389 | 18/1378
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 4/1389 | 14/1378
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 7/1389 | 11/1378
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7/1389 | 3/1378
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 4/1389 | 6/1378
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 6/1389 | 2/1378
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 6/1389 | 5/1378
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0/1389 | 4/1378
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 2/1389 | 4/1378
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 4/1389 | 3/1378
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1/1389 | 3/1378
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 3/1389 | 3/1378
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0/1389 | 2/1378
Respiratory Arrest (Respiratory, thoracic and mediastinal disorders) | 1/1389 | 2/1378
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0/1389 | 2/1378
Bronchitis Chronic (Respiratory, thoracic and mediastinal disorders) | 2/1389 | 1/1378
Foreign Body Aspiration (Respiratory, thoracic and mediastinal disorders) | 2/1389 | 0/1378
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2/1389 | 0/1378
Pulmonary Congestion (Respiratory, thoracic and mediastinal disorders) | 2/1389 | 0/1378
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 2/1389 | 0/1378
Asthma (Respiratory, thoracic and mediastinal disorders) | 0/1389 | 1/1378
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0/1389 | 1/1378
Bronchial Fistula (Respiratory, thoracic and mediastinal disorders) | 0/1389 | 1/1378
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 0/1389 | 1/1378
Lung Consolidation (Respiratory, thoracic and mediastinal disorders) | 0/1389 | 1/1378
Pulmonary Fibrosis (Respiratory, thoracic and mediastinal disorders) | 1/1389 | 1/1378
Respiratory Acidosis (Respiratory, thoracic and mediastinal disorders) | 0/1389 | 1/1378
Sleep Apnoea Syndrome (Respiratory, thoracic and mediastinal disorders) | 1/1389 | 1/1378
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0/1389 | 1/1378
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1/1389 | 0/1378
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1/1389 | 0/1378
Cough (Respiratory, thoracic and mediastinal disorders) | 1/1389 | 0/1378
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 1/1389 | 0/1378
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1/1389 | 0/1378
Lung Infiltration (Respiratory, thoracic and mediastinal disorders) | 1/1389 | 0/1378
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1/1389 | 0/1378
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1/1389 | 0/1378
Pulmonary Necrosis (Respiratory, thoracic and mediastinal disorders) | 1/1389 | 0/1378
Wegener's Granulomatosis (Respiratory, thoracic and mediastinal disorders) | 1/1389 | 0/1378
Skin Ulcer (Skin and subcutaneous tissue disorders) | 11/1389 | 10/1378
Skin Necrosis (Skin and subcutaneous tissue disorders) | 2/1389 | 2/1378
Diabetic Ulcer (Skin and subcutaneous tissue disorders) | 2/1389 | 1/1378
Cutaneous Vasculitis (Skin and subcutaneous tissue disorders) | 0/1389 | 1/1378
Dermatitis Exfoliative (Skin and subcutaneous tissue disorders) | 0/1389 | 1/1378
Ingrowing Nail (Skin and subcutaneous tissue disorders) | 0/1389 | 1/1378
Pemphigus (Skin and subcutaneous tissue disorders) | 0/1389 | 1/1378
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 1/1389 | 0/1378
Dry Gangrene (Skin and subcutaneous tissue disorders) | 1/1389 | 0/1378
Nail Discolouration (Skin and subcutaneous tissue disorders) | 1/1389 | 0/1378
Refusal Of Treatment By Patient (Vascular disorders) | 0/1389 | 1/1378
Arterial Bypass Operation (Vascular disorders) | 0/1389 | 1/1378
Catheter Placement (Vascular disorders) | 0/1389 | 1/1378
Chemotherapy Neurotoxicity Attenuation (Vascular disorders) | 1/1389 | 0/1378
Parathyroidectomy (Vascular disorders) | 1/1389 | 0/1378
Peripheral Ischaemia (Vascular disorders) | 24/1389 | 14/1378
Hypotension (Vascular disorders) | 14/1389 | 20/1378
Peripheral Arterial Occlusive Disease (Vascular disorders) | 15/1389 | 10/1378
Hypertension (Vascular disorders) | 11/1389 | 11/1378
Peripheral Vascular Disorder (Vascular disorders) | 5/1389 | 10/1378
Hypertensive Crisis (Vascular disorders) | 8/1389 | 6/1378
Extremity Necrosis (Vascular disorders) | 7/1389 | 4/1378
Arteriosclerosis (Vascular disorders) | 5/1389 | 6/1378
Haematoma (Vascular disorders) | 6/1389 | 3/1378
Aortic Aneurysm (Vascular disorders) | 2/1389 | 4/1378
Arteritis (Vascular disorders) | 0/1389 | 4/1378
Aortic Aneurysm Rupture (Vascular disorders) | 1/1389 | 3/1378
Cardiovascular Insufficiency (Vascular disorders) | 1/1389 | 3/1378
Deep Vein Thrombosis (Vascular disorders) | 2/1389 | 3/1378
Femoral Artery Occlusion (Vascular disorders) | 0/1389 | 3/1378
Shock (Vascular disorders) | 1/1389 | 3/1378
Venous Stenosis (Vascular disorders) | 3/1389 | 3/1378
Aortic Stenosis (Vascular disorders) | 2/1389 | 2/1378
Circulatory Collapse (Vascular disorders) | 2/1389 | 2/1378
Intermittent Claudication (Vascular disorders) | 1/1389 | 2/1378
Peripheral Artery Aneurysm (Vascular disorders) | 0/1389 | 2/1378
Steal Syndrome (Vascular disorders) | 1/1389 | 2/1378
Superior Vena Caval Stenosis (Vascular disorders) | 1/1389 | 2/1378
Vena Cava Thrombosis (Vascular disorders) | 1/1389 | 2/1378
Venous Occlusion (Vascular disorders) | 0/1389 | 2/1378
Arterial Stenosis Limb (Vascular disorders) | 2/1389 | 1/1378
Femoral Arterial Stenosis (Vascular disorders) | 2/1389 | 1/1378
Hypovolaemic Shock (Vascular disorders) | 2/1389 | 0/1378
Iliac Artery Stenosis (Vascular disorders) | 2/1389 | 1/1378
Subclavian Artery Stenosis (Vascular disorders) | 2/1389 | 0/1378
Aneurysm (Vascular disorders) | 0/1389 | 1/1378
Aneurysm Ruptured (Vascular disorders) | 0/1389 | 1/1378
Aortic Dissection (Vascular disorders) | 0/1389 | 1/1378
Arterial Disorder (Vascular disorders) | 0/1389 | 1/1378
Arterial Stenosis (Vascular disorders) | 0/1389 | 1/1378
Arterial Thrombosis Limb (Vascular disorders) | 1/1389 | 1/1378
Arteriosclerosis Obliterans (Vascular disorders) | 1/1389 | 1/1378
Blue Toe Syndrome (Vascular disorders) | 0/1389 | 1/1378
Diabetic Vascular Disorder (Vascular disorders) | 0/1389 | 1/1378
Hypertensive Emergency (Vascular disorders) | 0/1389 | 1/1378
Iliac Artery Occlusion (Vascular disorders) | 0/1389 | 1/1378
Ischaemic Limb Pain (Vascular disorders) | 0/1389 | 1/1378
Lymphoedema (Vascular disorders) | 0/1389 | 1/1378
Necrosis Ischaemic (Vascular disorders) | 1/1389 | 1/1378
Poor Peripheral Circulation (Vascular disorders) | 1/1389 | 1/1378
Shock Haemorrhagic (Vascular disorders) | 1/1389 | 1/1378
Subclavian Vein Thrombosis (Vascular disorders) | 0/1389 | 1/1378
Thrombophlebitis (Vascular disorders) | 0/1389 | 1/1378
Vascular Calcification (Vascular disorders) | 0/1389 | 1/1378
Venous Aneurysm (Vascular disorders) | 0/1389 | 1/1378
Aortic Occlusion (Vascular disorders) | 1/1389 | 0/1378
Arterial Insufficiency (Vascular disorders) | 1/1389 | 0/1378
Lymphocele (Vascular disorders) | 1/1389 | 0/1378
Orthostatic Hypotension (Vascular disorders) | 1/1389 | 0/1378
Peripheral Embolism (Vascular disorders) | 1/1389 | 0/1378
Secondary Hypertension (Vascular disorders) | 1/1389 | 0/1378
Thrombophlebitis Superficial (Vascular disorders) | 1/1389 | 0/1378
Thrombosis (Vascular disorders) | 1/1389 | 0/1378
Vasculitis (Vascular disorders) | 1/1389 | 0/1378
Venous Thrombosis (Vascular disorders) | 1/1389 | 0/1378
Venous Thrombosis Limb (Vascular disorders) | 1/1389 | 0/1378
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rosuvastatin 10mg (N=1389) | Placebo (N=1378)
Anaemia (Blood and lymphatic system disorders) | 81 | 62
Atrial Fibrillation (Cardiac disorders) | 70 | 59
Diarrhoea (Gastrointestinal disorders) | 202 | 188
Vomiting (Gastrointestinal disorders) | 112 | 127
Nausea (Gastrointestinal disorders) | 121 | 97
Constipation (Gastrointestinal disorders) | 82 | 80
Abdominal Pain (Gastrointestinal disorders) | 80 | 74
Bronchitis (Infections and infestations) | 129 | 133
Nasopharyngitis (Infections and infestations) | 127 | 116
Urinary Tract Infection (Infections and infestations) | 92 | 83
Arteriovenous Fistula Site Complication (Injury, poisoning and procedural complications) | 131 | 131
Haemodialysis-Induced Symptom (Injury, poisoning and procedural complications) | 79 | 78
Procedural Hypotension (Injury, poisoning and procedural complications) | 76 | 75
Arthralgia (Musculoskeletal and connective tissue disorders) | 110 | 93
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 90 | 101
Back Pain (Musculoskeletal and connective tissue disorders) | 97 | 92
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 97 | 81
Headache (Nervous system disorders) | 109 | 112
Insomnia (Psychiatric disorders) | 68 | 77
Cough (Respiratory, thoracic and mediastinal disorders) | 120 | 125
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 102 | 99
Pruritus (Skin and subcutaneous tissue disorders) | 83 | 69
Hypotension (Vascular disorders) | 115 | 109
Hypertension (Vascular disorders) | 102 | 92

LIMITATIONS AND CAVEATS:
The endpoints were originally intended to be time to event endpoints, however we are unable to report the data as intended due to the nature of time to event endpoints. Therefore we have reported the number of participants who reached the event.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No